CLINICAL TRIAL: NCT04528836
Title: A Phase 1/1B First-in-Human Study of the SHP2 Inhibitor BBP-398 (Formerly Known as IACS-15509) in Patients With Advanced Solid Tumors
Brief Title: First-in-Human Study of the SHP2 Inhibitor BBP-398 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Navire Pharma Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAV-1001
Record Dates: First submitted 2020-07-27; First posted 2020-08-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Tumor, Solid
Keywords: Cancer; MAPK-pathway alterations
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Oral capsules taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 28 days in duration with BBP-398 administered, once daily (QD).
  Interventions: Drug: BBP-398 (Formerly known as IACS-15509)
- Dose Expansion (Experimental): Oral capsules administered at MTD/RP2D defined dose. Each treatment cycle will be 28 days in duration with BBP-398 administered, once daily (QD)
  * Cohort A: Advanced or metastatic KRAS mutant solid tumor
  * Cohort B: Advanced solid tumor with NF1 loss-of-function (LOF) or metastatic BRAF class II/III mutant solid tumor
  Interventions: Drug: BBP-398 (Formerly known as IACS-15509)

INTERVENTIONS:
Drug: BBP-398 (Formerly known as IACS-15509) — oral capsules

SUMMARY:
A first-in-human study to evaluate the safety, tolerability and maximum tolerated dose (MTD) and establish the recommended phase 2 dose (RP2D) of BBP-398, a SHP2 inhibitor, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The first-in-human (FIH) study of BBP-398 will be an open-label, sequential-cohort, non-randomized, Phase 1/1B study utilizing BOIN dose escalation followed by an expansion phase in patients with MAPK pathway- or RTK-driven advanced solid tumors. The primary objective is to determine safety and tolerability of BBP-398, the MTD and RP2D. The secondary objectives are to assess the pharmacokinetic (PK) and pharmacodynamic (PD) profile, preliminary anti-tumor activity, objective response rate (ORR, complete response + partial response rate) and the duration of response (DoR) of BBP-398. The exploratory objective is to assess predictive biomarkers of response.

ELIGIBILITY:
Key Inclusion Criteria

* Male and non-pregnant females >18 years old.
* Patients must have a diagnosis of advanced (primary or recurrent) or metastatic solid tumor with MAPK-pathway alterations as assessed by clinically validated and/or FDA-approved molecular diagnostic and no available standard of care or curative therapies (MAPK-pathway alterations include, for example KRASG12C mutant, EGFR-mutant).
* Dose expansion only: Patients with specific genomically defined tumor types will be recruited.
* Patients must have measurable disease by RECIST v1.1.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
* Patients must have adequate organ function.
* Patients must have the ability to understand and the willingness to sign a written informed consent document prior to the initiation of the study and any study procedures.
* Patients must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures.

Key Exclusion Criteria

* Patients with known active Hepatitis B, Hepatitis C infection, or HIV infection.
* Patients with a history of CVA, myocardial infarction or unstable angina within the previous 6 months before starting therapy.
* Patients with clinically significant cardiac disease.
* Patients with tumors harboring known activating mutations.
* Patients with a known additional malignancy that is progressing or requires active treatment.
* Patients with known central nervous system (CNS) tumors.
* Patients with known active CNS metastases and/or carcinomatous meningitis.
* Patients who have previously received a SHP2 inhibitor.
* Patients with inability to swallow oral medications or with gastrointestinal illness that would preclude the absorption of an oral agent.
* Patients on dialysis.
* Patients with a life expectancy of ≤12 weeks after the start of IP according to the investigator's judgement.
* Patients with known intolerance/hypersensitivity to BBP-398 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) and establish the RP2D of BBP-398. | Completion of 1 Cycle ( 28 days)
  The MTD will be based on DLT.

SECONDARY OUTCOMES:
Determination of anti-tumor activity of BBP-398 | After 1 dose of BBP-398
  Anti-tumor activity will be defined by objective response rate (ORR2, complete response + partial response rate) and duration of response (DOR3)
Maximum observed plasma concentration (Cmax) of BBP-398 | Approximately 6 weeks
  Maximum plasma concentration of BBP-398 after single and multiple dose administration of BBP-398
Time to reach Cmax (Tmax) of BBP-398 | Approximately 6 weeks
  The amount of time to reach Cmax after single and multiple dose administration of BBP-398
Terminal half-life (t1/2) of BBP-398 | Approximately 6 weeks
  Terminal half-life (t1/2) after single and multiple dose administration of BBP-398
Area under the plasma concentration-time curve (AUC) of BBP-398 | Approximately 6 weeks
  Area under the plasma concentration versus time curve after single and multiple dose administration of BBP-398

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Scripps MD Anderson Cancer Center, La Jolla, California
  - UC Irvine Health, Orange, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington